CLINICAL TRIAL: NCT05854212
Title: Behavioral Economics to Implement a Traffic Light Nutrition Ranking System in a Network of Food Pantries
Brief Title: Behavioral Economics to Implement Nutrition Ranking in Food Pantries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023p001207
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity; Dietary Quality; Behavioral Economics; Implementation Science

STUDY DESIGN:
Intervention Model Description: Food agencies will be randomized to one of two interfaces on the online food bank ordering platform.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be automatically obtained from the food bank database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral economics-enhanced user interface (Experimental): Food agencies will see the behavioral economics (BE)-enhanced interface by default; food items will be sorted with green-labeled items listed first, followed by yellow, then red. If users search for a specific item type (e.g., chicken) the results returned for that item type will also be sorted so that green-labeled items are listed first. At any time during the ordering episode, users will have the option to switch from the BE-enhanced default to an alternate sorting or filtering choice, such as alphabetical or cost. Users will be shown the percent of items (by weight) that are labeled green in a prominent location on the ordering screen. The percent green-labeled items in the order will appear alongside messaging reporting the average percent green-labeled items ordered by GBFB pantries that rank in the top 10% based on this metric. Agencies will receive monthly emails from GBFB about SWAP, describing why common items receive certain SWAP rankings (e.g., item is yellow vs green).
  Interventions: Behavioral: Behavioral economics-enhanced user interface
- Usual user interface (No Intervention): When agency staff log on to the food bank platform, by default, foods are listed in alphabetical order. If they wish, users can change how items are sorted or filtered using pull-down menus and check-boxes, including the ability to have items sorted or filtered based on traffic light labels. As orders are created, an information section at the top of the page is updated with details on the order weight and cost. Agencies will not receive emails about SWAP.

INTERVENTIONS:
Behavioral: Behavioral economics-enhanced user interface — The intervention changes the ordering platform visible to food agencies using behavioral economics strategies to promote healthier food choices.
  Arms: Behavioral economics-enhanced user interface

SUMMARY:
The goal of this randomized controlled trial is to test whether using behavioral economic strategies to promote healthy food choices on a food bank's online ordering platform increases the use of the traffic light nutrition ranking system and increases healthier food selections by the food agencies (e.g., food pantries) who use the food bank.

DETAILED DESCRIPTION:
This study will use behavioral economic strategies to promote utilization of traffic-light nutrition ranking in the Greater Boston Food Bank (GBFB) order system to improve the dietary quality of food ordered by GBFB agencies. Supporting Wellness at Pantries (SWAP) is a program to guide both traffic light labeling for use on ordering platforms and pantry shelves, as well as food pantry layout to inform clients and encourage healthy food choice.This study is a collaboration with the Greater Boston Food Bank (GBFB) to test BE strategies (choice architecture, framing, social norms) for implementation of an evidence-based intervention (traffic light nutrition ranking, SWAP). We will determine if behavioral economic interventions on the GBFB online ordering platform increase agencies' use of traffic light nutrition labels when placing orders and increases their healthy food orders. We will conduct a 12-month randomized controlled trial comparing agencies' ordering experiences and outcomes with the current user interface (control) to a "SWAP-enhanced" user interface (intervention). All GBFB partner agencies will be randomized to see either the control or intervention interfaces when they log on to ShopGBFB, GBFB's online food ordering platform. In addition, intervention group agencies will receive monthly emails from GBFB about SWAP labeling, such as why common items receive certain rankings (e.g., canned green beans will have a yellow label if there is added sodium) and common misunderstandings people have about SWAP labels (e.g., explaining why all chicken items do not get the same SWAP ranking). At the end of 12 months, agency staff will complete a survey about their online ordering experiences at GBFB. In the next phase, the SWAP-enhanced ShopGBFB interface will be updated, adapted, and implemented for all 364 agencies that place orders. Agency ordering outcomes will be monitored for 12 additional months.

ELIGIBILITY:
Inclusion Criteria:

* Food agencies that order food from the Greater Boston Food Bank (GBFB) online ordering platform.

Exclusion Criteria:

* Food agencies that do not order food from the GBFB online platform within 2 months of the start of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Healthy food agency orders from the food bank | 12 months
  This will be the change from baseline to 12 months in the percentage of foods ordered (by weight) that have green labels.

SECONDARY OUTCOMES:
Proportion of agencies that ever used the traffic light label sorting or filtering when ordering from the food bank | 12 months
  This outcome will be the proportion of agencies in the intervention vs. control group that report using the traffic-light sorting/filtering when making orders during the 12 month intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No